CLINICAL TRIAL: NCT00404885
Title: A Double-Masked, Placebo-Controlled, Parallel-Group, Multi-Center, Dose-Ranging Study With an Optional Extension to Assess the Efficacy and Safety of LX211 as Therapy in Subjects With Active Sight Threatening, Non-infectious Anterior Uveitis
Brief Title: A Multi-center Study to Assess the Efficacy and Safety of LX211 in Active Non-infectious Anterior Uveitis
Acronym: LUMINATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lux Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX211-03-UV; EudraCT No: 2006-006545-13
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Uveitis, Anterior; Panuveitis
Keywords: uveitis; calcineurin; inflammation
MeSH Terms: conditions — Uveitis, Anterior; Panuveitis; Uveitis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- LX211, 0.2 mg/kg (Active Comparator)
  Interventions: Drug: LX211
- LX211, 0.4 mg/kg (Active Comparator)
  Interventions: Drug: LX211
- LX211, 0.6 mg/kg (Active Comparator)
  Interventions: Drug: LX211

INTERVENTIONS:
Drug: Placebo — PO BID
  Arms: Placebo
Drug: LX211 — 0.2 mg/kg, twice a day (BID)
  Arms: LX211, 0.2 mg/kg
Drug: LX211 — 0.4 mg/kg, twice a day (BID)
  Arms: LX211, 0.4 mg/kg
Drug: LX211 — 0.6 mg/kg, twice a day (BID)
  Arms: LX211, 0.6 mg/kg

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of LX211 as therapy in subjects with active non-infectious anterior uveitis

ELIGIBILITY:
Inclusion Criteria:

* Documented history of non-infectious anterior, anterior and intermediate- or panuveitis
* Currently uncontrolled uveitis for a minimum of 2 weeks despite use of oral and/or topical corticosteroid,or subjects who are intolerant of local corticosteroid therapy due to the development of an ocular hypertensive response or subjects for whom oral corticosteroid is contraindicated.
* Grade of 2+ or higher for anterior chamber cells at time of enrollment
* Considered by the investigator to require corticosteroid-sparing therapy.
* Subjects not planning to undergo elective ocular surgery during the study

Exclusion Criteria:

* Uveitis of infectious etiology
* Presence of an ocular toxoplasmosis scar
* An immune suppression regimen that includes an alkylating agent within the previous 90 days

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
anterior chamber cells | 16 and 24 weeks

SECONDARY OUTCOMES:
BCVA | 24 weeks
macular thickness | 16 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Anglade, M.D., Study Chair — Chief Medical Officer
Locations (30):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - University of Illinois - Chicago, Chicago, Illinois
  - Wilmer Eye Institute, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Massachusetts Eye Research and Surgery Institute, Cambridge, Massachusetts
  - Associated Retinal Consultants, PC, Grand Rapids, Michigan
  - Tauber Eye Center, Kansas City, Missouri
  - New York Eye & Ear Hospital, New York, New York
  - Duke University Eye Center, Erwin Road, Durham, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - Brian B. Berger, MD, P.A., Austin, Texas
  - Retina & Uveitis Consultants of Texas, San Antonio, Texas
  - Viginia Eye Consultants, Norfolk, Virginia
- Austria (2):
  - Universitätsklinik für Augenheilkunde, Salzburg
  - Klinik für Augenheilkunde, Dept. of Ophthalmology, Vienna
- McGill University Health Center, Montreal, Quebec, Canada
- Hôpital Pitié Salpétrière, Service d'Ophtalmologie, Paris, France
- Germany (4):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Augenklinik der Universität Heidelberg, Heidelberg
  - St. Franziskus-Hospital, Münster
  - Universitätsklinikum Tübingen, Tübingen
- India (6):
  - L V Prasad Eye Institute, Hyderabaad, Andhra Pradesh
  - Aravind Eye Hospitals and Postgraduate Institute of Ophthalmology, Madurai, Tamil Nadu
  - Vittala International Institute of Ophthalmology, Bangalore
  - Advanced Eye Centre, Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh
  - Aravind Eye Hospital, Uvea Clinic, Coimbatore
  - Aditya Jyot Eye Hospital Pvt Ltd, Mumbai
- United Kingdom (2):
  - Bristol Eye Hospital and University of Bristol, Bristol
  - Royal Liverpool University Hospital, Liverpool

REFERENCES:
- See also: Related Info — http://www.luxbio.com